CLINICAL TRIAL: NCT04936958
Title: RETR(Osteomyelitis)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 405
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-05

CONDITIONS: Osteomyelitis
Keywords: hematogenous; bone substitute
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had an osteomyelitis since 2017
  Interventions: Other: patients having had an osteomyelitis since 2017

INTERVENTIONS:
Other: patients having had an osteomyelitis since 2017 — description of osteomyelitis and their management

SUMMARY:
This is a retrospective study describing the management of osteomyelitis in a referece center, with success and failures.

DETAILED DESCRIPTION:
Chronic osteomyelitis is a serious osteoarticular infection that most often occurs in the long bones (tibia, femur, humerus), responsible for significant morbidity with the risk of fracture and amputation. It is caused by the presence of bacteria in the bone marrow, sometimes responsible for an intraosseous abscess. Chronic osteomyelitis can have a hematogenous or more often exogenous origin, after trauma or surgery.

Despite the progress made in both antibiotics and surgical treatment, the probability of failure of this treatment (infectious recurrence) is of the order of 20%, and has unfortunately remained stable for more than 20 years.

An innovative treatment, Cerament-G (BONESUPPORT AB Laboratory, Sweden), a synthetic bone substitute composed of hydroxyapatite, calcium sulphate, and gentamicin (CE marking), fills the "dead space" which is formed during surgery, prevents this cavity filled with blood from becoming infected, and promotes the regeneration of the bone within this space, limiting the risk of fracture in the medium and long term. It also locally delivers very high doses of gentamicin for several weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with osteomyelitis between 2017 and 2021

Exclusion Criteria:

* Patients who objected to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who presented with osteomyelitis between 2017 and 2021 managed at the CRIOAc Lyon
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
rate of osteomyelitis in BJI | between 2017 and 2021
  proportion of patients having had an osteomyelitis
site of osteomyelitis | between 2017 and 2021
  localisation
bone defect size | between 2017 and 2021
  dimension of the bone defect size
type of osteomyelitis | between 2017 and 2021
  hematogenous or after a trauma or after a surgery
rate of bacteria involved in osteomyelitis | between 2017 and 2021
  description of bacteria responsible for osteomyelitis
Description of patients | between 2017 and 2021
  comorbidities, age
Description of the follow up of the patients | between 2017 and 2021
  duration of the follow up of patients
description of patients : medical treatment | between 2017 and 2021
  description and duration of antibiotics
Description of patients : surgical treatment | between 2017 and 2021
  description of surgery performed
rate of patient treated with CERAMENT | between 2017 and 2021
  proportion of patients having had CERAMENT
rate of treatment failure | between 2017 and 2021
  treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/